CLINICAL TRIAL: NCT05114499
Title: Efficacy and Safety of Donepezil and Sodium Oligomannate in Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021LSK-328
Record Dates: First submitted 2021-11-05; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; GV-971

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Donepezil monotherapy group: Donepezil 5mg qd
  Interventions: Drug: Donepezil
- GV-971 monotherapy group: GV-971 450mg bid
  Interventions: Drug: GV-971
- Donepezil combined with GV-971 group: Donepezil 5mg qd+GV-971 450mg bid
  Interventions: Drug: Donepezil; Drug: GV-971

INTERVENTIONS:
Drug: Donepezil — Donepezil 5mg qd
  Groups: Donepezil combined with GV-971 group; Donepezil monotherapy group
Drug: GV-971 — GV-971 450mg bid
  Groups: Donepezil combined with GV-971 group; GV-971 monotherapy group

SUMMARY:
Alzheimer's disease (AD) is the main cause of dementia. At present, AD is incurable. Cholinesterase inhibitors, especially donepezil, are the first choice for mild and moderate AD. Sodium oligomannate (GV-971) is a marine-derived oligosaccharide. It is proposed that it can reconstitute the gut microbiota, and inhibit neuroinflammation in the brain as observed in animal models. It reduces Aβ deposition in the brain of Aβ-transgenic mice. The reduction in both Aβ deposition and neuroinflammation may synergistically contribute to the improvement of cognitive impairment and delay the progress of the disease. The State Food and Drug Administration of China (SFDA) approved it for the treatment of mild to moderate AD in 2019. Due to the different mechanism of cholinesterase inhibitor and GV-971, theoretically, they may synergistically improve cognitive function and delay disease progression. They are also used in patients with AD, but there is a lack of data on their effectiveness and safety. Therefore, the purpose of this observational study is to compare the efficacy and safety of donepezil and GV-971 monotherapy and combination therapy in patients with mild and moderate AD, which is of great significance for guiding the treatment of mild and moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* age of 50-85 years old , either sex;
* met the diagnostic criteria for suspected AD;
* mild to moderate AD patients, that is, patients with 11 points ≤Mini-Mental State Examination(MMSE) total score ≤26 points
* total Hachinski ischemic scale (HIS) score ≤4 points;
* memory loss for at least 12 months, with a tendency of progressive deterioration;
* brain magnetic resonance imaging（MRI） scan suggesting a significant possibility of AD ;
* no obvious physical signs during nervous system examination;
* stable and reliable caregivers,
* elementary school or higher education level
* signed an informed consent form

Exclusion Criteria:

* previous nervous system diseases (including stroke, optic neuromyelitis, Parkinson's disease, epilepsy, etc.);
* mental illness according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition（DSM-IV), Text Revision criteria, including schizophrenia and other mental illness, bipolar disorder, and severe depression or paralysis;
* unstable or severe heart, lung, liver, kidney, or hematopoietic diseases;
* uncorrectable visual and auditory disorders that affected completing neuropsychological tests and scale assessments;
* simultaneous use of cholinesterase inhibitors or memantine.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be enrolled from our memory clinic and in-patients and should meet the the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) (1984) criteria for probable AD.The diagnosis of AD is mainly based on detail clinical history from caregivers, neuropsychological testing, and brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cognitive function | baseline, week 12, week 24, week 36
  the change of Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-cog) score from baseline at week 36